CLINICAL TRIAL: NCT05394766
Title: A Pragmatic RCT of Remote Patient Monitoring and Health Coaching vs. Usual Care for the Treatment of Hypertension
Brief Title: Remote Patient Monitoring and Health Coaching vs. Usual Care for the Treatment of Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Omada Health, Inc. (Industry)
Responsible Party: Principal Investigator, Steven Lin, Clinical Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65790
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Does not receive access to Omada Health program (No Intervention): Participants manage hypertension with usual care alone.
- Receives access to Omada Health program (Experimental): In addition to usual care, participants will gain access to the Omada Program, an online program that offers lifestyle self-management support for hypertension. Participants will be assigned a health coach and a hypertension specialist via Omada's secure app. Participants will receive hypertension education and resources and communicate with their care team through asynchronous, in-app messaging features. Participants will receive digital tools that connect with the Omada app to help track their food intake, physical activity, and blood pressure (BP). Participants who also have diabetes will receive a digital blood glucose meter and/or a continuous glucose monitor as well. The care team will support patients with lifestyle self-management support, adherence to their current medication regimen, improved BP control, and use of monitors for self-management of their BP and/or blood glucose values.
  Interventions: Other: Omada Hypertension Program

INTERVENTIONS:
Other: Omada Hypertension Program — The Omada Program: an online program that offers comprehensive lifestyle self-management support for hypertension.
  Arms: Receives access to Omada Health program

SUMMARY:
High blood pressure, also known as hypertension, affects nearly half of all Americans and increases the risk for heart disease and stroke. Only about half of people with high blood pressure have it under control. New methods to control blood pressure are needed to reduce heart attack and stroke rates. The purpose of this study is to test whether a digital program that includes personalized health coaching and remote patient monitoring with a connected blood pressure cuff, all delivered on a smartphone or website, can improve blood pressure control compared with usual care among patients with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* 18+ years of age
* English-speaking
* Receives primary care at Stanford Primary Care

Exclusion Criteria:

* <18 years of age
* Primary language not English
* Active or prior enrollment in Omada Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in systolic blood pressure at 1-year | Baseline, 1 year

SECONDARY OUTCOMES:
Mean change from baseline in A1c at 1-year | Baseline, 1 year
Mean change from baseline in weight at 1-year | Baseline, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No